CLINICAL TRIAL: NCT01317862
Title: A Comparison of Transcervical Foley Catheter and Prostaglandins for Induction of Labor at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCB_PG_01
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Failed Induction of Labor
Keywords: labor induction, transcervical foley catheter, prostaglandin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcervical foley catheter (Active Comparator)
  Interventions: Device: Transcervical foley catheter, Prostaglandins
- Prostaglandins (Active Comparator)
  Interventions: Device: Transcervical foley catheter, Prostaglandins

INTERVENTIONS:
Device: Transcervical foley catheter, Prostaglandins — 16 French foley catheter 10mg dinoprostone vaginal insert

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of transcervical foley catheter as compared to prostaglandins for preinduction cervical ripening and labor induction in term nulliparous women with unfavorable cervix.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* nulliparous women
* gestational age >= 37.0 weeks
* Bishop score <= 5
* intact amniotic membrane
* abscence of labor
* live fetus with vertex presentation
* no previous uterine surgical procedure

Exclusion Criteria:

* major congenital anomaly

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Successful labor induction | Twelve hours of initiating oxytocin on the fist day of induction
  Successful labor induction is defined as an ability to achieve the active phase of labor corresponding to a cervical dilatation of >=4cm.

SECONDARY OUTCOMES:
Cervical change in the bishop scores and cervical lengths induced by transcervical foley catheter and prostaglandins | When transcervical foley catheter or prostagladins was removed befor adminitoring oxytocin
  1. Cervical change based on the bishop score and cervical length induced by cervical ripening method(foley catheter balloon vs prostaglandin)
  2. Incidence of cesarean delivery
  3. Vaginal delivery with 24 hours of starting of induction
  4. The interval from start of oxytocin to delivery
  5. Incidence of admission to neonatal intensive care unit and uterine tachysystole
  6. Pain score by the type of ripening method

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Hoon Park, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Obstetrics and Gynecology Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264